CLINICAL TRIAL: NCT06472453
Title: Prospective Comparative Evaluation of Alveolar Ridge Preservation: Mixing Allograft With Xenograft VS. Allograft Alone in Atraumatic Extraction Sockets
Brief Title: Vallomix Socket Preservation Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HP-00110704; SAP# 101-080 (Other Grant/Funding Number: Geistlich Pharma North America Inc.)
Record Dates: First submitted 2024-05-28; First posted 2024-06-25 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Alveolar Ridge Augmentation
MeSH Terms: interventions — Transplantation, Homologous; Transplantation, Heterologous

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Alveolar ridge preservation with Allograft/Xenograft group (Experimental): The patients in both groups will go through the same treatment but with two different bone grafting materials depending on the assigned group. The patients in this group will have alveolar ridge preservation with the mixture of demineralized cortical allograft vallos®f and xenograft bone substitute called Bio-Oss®.
  Interventions: Device: Allograft/Xenograft
- Alveolar ridge preservation with Allograft group (Active Comparator): The patients in both groups will go through the same treatment but with two different bone grafting materials depending on the assigned group. The patients in this group will have alveolar ridge preservation with mineralized cortico-cancellous bone substitute called vallos®.
  Interventions: Device: Allograft

INTERVENTIONS:
Device: Allograft/Xenograft — Alveolar ridge preservation of a single extraction socket site with a mixture of demineralized cortical bone substitute vallos®" and xenograft Bio-Oss®.
  Arms: Alveolar ridge preservation with Allograft/Xenograft group
Device: Allograft — Alveolar ridge preservation of a single extraction socket site with vallos® (mineralized cortico-cancellous bone substitute)
  Arms: Alveolar ridge preservation with Allograft group

SUMMARY:
This research aims to compare the effectiveness of two bone grafting materials on preserving jawbone integrity after tooth extraction. Following extraction, the jawbone surrounding the removed tooth can shrink, affecting future implant placement. By placing a bone graft material in the extraction socket, we aim to maintain adequate jawbone space for future implants. This study compares how well the mixture of vallos®f (human source bone) and Bio-Oss (animal source bone) [test], and vallos® only [control] grafting materials work.

Participants with at least one tooth planned for extraction and subsequent implant placement are sought for this study. Participants will be randomly assigned to either the mixture of vallos®f and Bio-Oss (test) group or the vallos® only (control) group.

Throughout the approximately 2-year study duration, participants will undergo oral exams, x-rays, surgical procedures, and follow-up visits. All participants will undergo routine tooth extraction, bone graft material placement, and dental implant placement. After the crown is placed on the implant, participants will attend follow-up visits.

Participation in the study is voluntary, and the alternative is to continue routine dental care. Risks include minor discomfort from procedures such as tooth extraction and implant placement. The major benefit of participation in the study is the preservation of jaw dimensions following extraction, which will simplify the placement of a dental implant.

ELIGIBILITY:
Inclusion criteria:

1. Provision of informed consent
2. At least 18 years old
3. In need of one posterior tooth (premolar or molar), excluding third molar molars, planned for extraction and replacement with a dental implant
4. Type I or II extraction socket/ ridge identified at the time of enrolment with cone-beam CT scan
5. At least one retained natural tooth adjacent to the study site

Exclusion criteria

1. Insufficient interocclusal or interdental space to allow for an implant- supported prosthesis
2. Previous interventions performed involving soft and/or bone grafting in the study site
3. Active treated caries
4. Uncontrolled periodontal disease present
5. Evidence of active periapical, radicular, or endodontic lesions on teeth adjacent to study site
6. History of recent extraction of an adjacent tooth (mesial and distal) to study site within 6 months of enrollment
7. Current smoker with self-reported history of more than 10 cigarettes or equivalent per day
8. Self-reported use of smokeless tobacco or e-cigarette
9. Self-reported history of current alcohol or drug abuse
10. Systemic or local disease or condition that would compromise bone metabolism, post-operative healing and/or osseointegration e.g. uncontrolled diabetes with self-reported most recent HbA1c > 8.0 within last six-month
11. Systemic corticosteroids or any other medication that would influence bone metabolism, post-operative healing, and/or osseointegration

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-01-13 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Three-dimensional hard and soft tissue change using CBCT/ intraoral scan | Over the course of the study (From the time of study enrollment Alveolar Ridge Preservation [Visit 2] to 1-year post implant-supported crown delivery [Visit 11]).
  Evaluate the efficacies of Alveolar Ridge Preservation in three-dimensional ridge hard and soft tissue change in volumetric and linear measurement using CBCT and intraoral scan over time

SECONDARY OUTCOMES:
Comparison of implant positions of digital planning based on the CBCT scan before and after Alveolar Ridge Preservation will be compared. | 4-5 months (Before Alveolar Ridge Preservation/ Enrollment [Visit 2] to 4-month follow-up [Visit 7])
  Evaluate the efficacies of Alveolar Ridge Preservation in achieving intended implant placement. The digital planning on the CBCT before and after the e-extraction digital planning
Histomorphometric analysis of the bone harvested from the grafted site | 5 months (At the time of implant placement [Visit 8])
  Evaluate the bone harvested from the re-grafted site for new bone formation/remaining graft residuals at the time of implant placement (Visit 8) by histomorphometric analysis

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland School of Dentistry, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No